CLINICAL TRIAL: NCT05806138
Title: A Randomized Controlled Trial of the Soluble Guanylate Cyclase Stimulator Vericiguat in Patients With Breast Cancer and Cancer Therapy-Related Cardiac Dysfunction (ELEVATE)
Brief Title: A Study of Vericiguat in People With Breast Cancer and Cancer Therapy-Related Cardiac Dysfunction
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-050
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Cardiac Dysfunction
Keywords: Vericiguat; Cancer Therapy-Related Cardiac Dysfunction (CTRCD); 23-050
MeSH Terms: conditions — Breast Neoplasms | interventions — vericiguat

STUDY DESIGN:
Intervention Model Description: This is a single center, open-label, randomized controlled trial of vericiguat in adult patients with breast cancer and Cancer Therapy-Related Cardiac Dysfunction (CTRCD).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vericiguat plus optimal medical therapy (Experimental): For patients randomized to vericiguat, a starting dose of 2.5mg will be initiated at the randomization visit. At pre-specified titration visits, subjects will be up-titrated to vericiguat 5mg and then to the target dose of vericiguat 10mg using titration criteria based on mean systolic blood pressure and evaluation for clinical symptoms. Vericiguat will be administered in the background of optimal medical therapy for cardiomyopathy/heart failure.
  Interventions: Drug: Vericiguat
- Optimal medical therapy (Active Comparator): For patients randomized to the control group, optimal medical therapy for cardiomyopathy/heart failure will be instituted throughout the study period.
  Interventions: Other: Optimal medical therapy

INTERVENTIONS:
Drug: Vericiguat — A starting dose of vericiguat 2.5 mg will be administered in-clinic at the Day 1 visit. Titration visits will occur on Days 14 and 28, with dose escalation to 5 mg and 10 mg.
  Arms: Vericiguat plus optimal medical therapy
Other: Optimal medical therapy — All subjects will be followed by a cardiologist throughout the study period and will receive optimal medical therapy for cardiomyopathy/heart failure following the ACCF/AHA and ESC Guidelines for the Management of Heart Failure recommendations, applied individually at the discretion of the treating investigator and in line with individual tolerability. This includes medications such as ßblockers, angiotensin converting enzyme inhibitors(ACEI), angiotensin receptor/neprilysin inhibitor (ARNI), angiotensin receptor blockers (ARB), and mineralocorticoid antagonists
  Arms: Optimal medical therapy

SUMMARY:
The purpose of this study is to find out if adding vericiguat to standard treatment for cancer therapy related cardiac dysfunction (CTRCD) is more effective than standard treatment alone. The addition of vericiguat to the usual treatment could help improve cardiac function, but it could also cause side effects. This study will help researchers find out whether this different treatment is better, the same as, or worse than the usual approach.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Biopsy proven breast cancer (stage I-IV)
* Cancer treatment related cardiac dysfunction (CTRCD), established by an absolute decrease in LVEF ≥ 10% from baseline/pre-treatment to < 53% and attributable to prior cardiotoxic cancer treatment, per the clinical investigator.
* Able to complete an acceptable baseline CPET, in the absence of high-risk ECG findings or other inappropriate response to exercise as determined by the PI, as defined by any of the following criteria:

  * Achieving a plateau oxygen consumption, concurrent with an increase in power output;
  * A respiratory exchange ratio ≥ 1.00;
  * Attainment of maximal predicted heart rate, as defined by a peak heart rate within 10bpm of the age predicted maximal heart rate (220 - Age[years]); or if on a beta-blocker, 164 - (age * 0.7)
  * Volitional exhaustion, as measured by a rating of perceived exertion (RPE) ≥ 18 on the BORG scale.
* Willing to use highly effective contraceptive measures if of child-bearing potential or if the patient's sexual partner is a woman of child-earing potential while receiving study drug and for 30 days after the last dose of study drug:

  * Female subjects should be using highly effective contraceptive measures, and must have a negative pregnancy test (within 6 months prior to study enrollment) and not be breast-feeding prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:
  * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
  * Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the postmenopausal range for the institution
  * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy, but not tubal ligation.
* Male subjects should be willing to use barrier contraception °Willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

* Systolic blood pressure < 90 mmHg
* Concurrent or anticipated use of a long-acting nitrate or NO donor (e.g., nitroglycerin, isosorbide dinitrate, isosorbide 5-mononitrate, pentaerythritol tetranitrate, nicorandil or transdermal NTG patch, or molsidomine).
* Concurrent or anticipated use of a phosphodiesterase inhibitor (e.g., vardenafil, tadalafil, or sildenafil).
* Cardiac comorbidity, including any of the following:

  * Hypertrophic cardiomyopathy, restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, cardiac sarcoidosis, or amyloid cardiomyopathy
  * Uncontrolled arrhythmia
  * Uncorrected congenital cardiac disease
  * Acute coronary syndrome, percutaneous coronary intervention, or coronary artery bypass graft surgery within 3 months prior to randomization.
  * Symptomatic carotid stenosis, or transient ischemic attack (TIA) or stroke within 3 months prior to randomization.
  * Cardiac transplantation
* Valvular heart disease requiring surgery or intervention
* Non-cardiac comorbidity, including any of the following:

  * eGFR < 15ml/min/1.73m^2 (based upon CKD-EPI, Cockroft-Gault, etc.)
  * Severe hepatic insufficiency (e.g., Child-Pugh C)
  * Severe pulmonary disease, such as requiring continuous home oxygen or interstitial lung disease
  * Other medical disorder or condition that in the opinion of the investigator would impair the subject's ability to participate or complete the study
* Subjects must not have any of the following absolute contraindications to cardiopulmonary exercise testing:

  * Acute myocardial infarction (within 30 days of any planned study procedures)
  * Unstable angina
  * Uncontrolled arrhythmias causing symptoms or hemodynamic compromise,
  * Symptomatic severe aortic stenosis
  * Recurrent syncope
  * Active endocarditis
  * Acute myocarditis or pericarditis
  * Acute pulmonary embolus or pulmonary infarction (within 3 months of any planned study procedures)
  * Thrombosis of lower extremities (within 3 months of any planned study procedures)
  * Suspected dissecting aneurysm
  * Uncontrolled asthma
  * Pulmonary edema
  * Room air desaturation at rest ≤85%
  * Respiratory failure
  * Acute noncardiopulmonary disorder that may affect exercise performance or be aggravated by exercise (i.e., infection, renal failure, thyrotoxicosis)
  * Mental impairment leading to inability to cooperate.
* Current alcohol and/or drug abuse
* Any other condition or intercurrent illness (e.g., symptomatic weight-bearing bone metastases or limited life expectancy < 6-9 months) that, in the opinion of the investigator, makes the participant a poor candidate for the trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Enrollment: 21 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2028-07-17 (Estimated); Study Completion 2028-07-17 (Estimated)

PRIMARY OUTCOMES:
change in CRF (measured by VO2peak) | up to 6 months
  For the primary analysis, intervention effect will be evaluated by comparing differences in mean VO2peak changes from baseline to month 6 between the investigational and control groups using the analysis of covariance approach (ANCOVA).

SECONDARY OUTCOMES:
CRF response rate | up to 6 months
  assessed by the number of participants with a change in VO2peak ≥ 1.32 ml O2 • kg-1 • min-1 (technical error of CRF measurement) from baseline to month 6. A change in VO2peak ≥ 1.32 ml O2 • kg-1 • min-1 will be considered a response, whereas a change in VO2peak < 1.32 ml O2 • kg-1 • min-1 will be considered a non-response.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Yu, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm